CLINICAL TRIAL: NCT02229942
Title: B-lymphocyte Depletion Using the Monoclonal Anti-CD20 Antibody Rituximab in Chronic Fatigue Syndrome/ Myalgic Encephalopathy (CFS/ME). A Multicentre, Randomized, Double-blind and Placebo Controlled Phase-III Study With Rituximab Induction and Maintenance Treatment.
Brief Title: B-lymphocyte Depletion Using Rituximab in Chronic Fatigue Syndrome/ Myalgic Encephalopathy (CFS/ME). A Randomized Phase-III Study.
Acronym: RituxME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: The Research Council of Norway (Other); Norwegian Department of Health and Social Affairs (Other Government); The Kavli Foundation (Unknown); Oslo University Hospital (Other); Trondheim University Hospital (Other); University Hospital of North Norway (Other); Sykehuset Telemark (Other Government); MEandYou Foundation (Unknown); The Norwegian ME association (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KTS-6-2014; 2014-000795-25 (EudraCT Number); 229035 (Other Grant/Funding Number: Research Council of Norway: project no 229035)
Record Dates: First submitted 2014-08-29; First posted 2014-09-03 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2018-02

CONDITIONS: Chronic Fatigue Syndrome/ Myalgic Encephalitis (CFS/ME)
Keywords: Chronic Fatigue Syndrome (CFS); Myalgic Encephalitis (ME); Rituximab; B-lymphocyte depletion; B-cell depletion
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Rituximab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab (Experimental): Rituximab induction (two infusions two weeks apart) and maintenance (infusions at 3, 6, 9 and 12 months)
  Interventions: Drug: Rituximab
- Placebo (Placebo Comparator): Saline (with added albumin), two infusions two weeks apart, followed by infusions at 3, 6, 9 and 12 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rituximab — Induction with two infusions two weeks apart, rituximab 500 mg/m2 (max 1000 mg).
  Maintenance with rituximab infusions (500 mg fixed dose) at 3, 6, 9 and 12 months.
  Other Names: Rituxan; Mabthera
  Arms: Rituximab
Drug: Placebo — Saline (NaCl 0,9%) added human albumin (Flexbumin) 0,4 mg/ml, two infusions two weeks apart. Maintenance infusions after 3,6, 9 and 12 months.
  Other Names: Saline
  Arms: Placebo

SUMMARY:
The hypothesis is that a subgroup of patients with Chronic Fatigue Syndrome/ Myalgic Encephalopathy (CFS/ME) have a chronically activated immune system and may benefit from B-lymphocyte treatment using the monoclonal anti-CD20 antibody rituximab with induction and maintenance treatment.

DETAILED DESCRIPTION:
We have published a case series of pilot patient observations with B-cell depletion in Chronic Fatigue Syndrome/ Myalgic Encephalopathy (CFS/ME) (Fluge and Mella, BMC Neurol, 2009). Subsequently, we published a small randomized and double-blind phase II study using rituximab induction two infusions two weeks apart (Fluge et al, Plos One, 2011).

We have completed an open label phase II study with 29 patients using rituximab induction and maintenance treatment (six rituximab infusions over 15 months, with follow-up for three years, unpublished).

We hypothesize that a subgroup of patients with Chronic Fatigue Syndrome/ Myalgic Encephalopathy (CFS/ME) have a chronically activated immune system involving B-lymphocytes, possibly a variant of an autoimmune disease, and that patients may benefit from B-cell depletion therapy.

Three substudies will be performed:

Endothelial function: assessment of Flow-Mediated Dilation and skin microcirculation at baseline and repeated during the time interval 17-21 months.

Cardiopulmonary exercise test for two following days: assessment at baseline and repeated during the time interval 17-21 months.

Gastrointestinal function: assessment at baseline and repeated during the time interval 17-21 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Chronic Fatigue Syndrome/ Myalgic Encephalopathy (CFS/ME) according to Canadian diagnostic criteria (Carruthers, 2003)
* Duration of CFS/ME disease 2-15 years. For patients with mild CFS/ME duration of disease must be 5-15 years.
* Mild, Mild/Moderate, Moderate, Moderate/Severe and Severe CFS/ME may be included
* Signed informed consent

Exclusion Criteria:

* Patients with fatigue, who do not comply with Canadian diagnostic criteria (2003)
* Duration of CFS/ME < 2 years or >15 years
* Patients with very severe CFS/ME
* Pregnancy or lactation.
* Previous malignant disease (except basal cell carcinoma in skin or uterine cervical dysplasia)
* Previous treatment with B-lymphocyte depleting therapeutic monoclonal antibodies, such as rituximab
* Previous long-term systemic immunosuppressive treatment, including drugs such as cyclosporine, azathioprine, mycophenolate mofetil, but except steroid treatment e.g. for obstructive lung disease or for other autoimmune diseases such as ulcerative colitis
* Severe endogenous depression
* Lack of ability to adhere to protocol
* Known multi-allergy with clinically assessed risk from rituximab infusion
* Reduced kidney function (serum creatinine > 1,5x upper normal level)
* Reduced liver function (serum bilirubin or transaminases > 1,5x upper normal level)
* Known HIV positivity, previous hepatitis B or hepatitis C
* Evidence of ongoing, active and clinically relevant infection
* Known immunodeficiency with risk from therapeutic B-cell depletion, such as hypogammaglobulinemia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Fatigue score, selfreported. | Course of Fatigue score during 24 months follow-up.
  Selfreported Fatigue score is registered every second week, as the mean score for the four symptoms: "Post-exertional malaise", "Fatigue", "Need for rest", "Daily functioning" (scale 0-6). Mean Fatigue scores for the time intervals 0-4, 4-8, 8-12, 12-16, 16-20, 20-24 months are recorded for each patient. These data are used for statistical analysis. The difference in course of Fatigue score during 24 months follow-up, between the rituximab and placebo groups, will constitute the primary endpoint.
  Overall response is recorded as the effect on CFS/ME symptoms during 24 months follow-up. The overall response is not predefined to a specific time interval, but is defined as mean Fatigue score at least 4.5 for at least 8 consecutive weeks for moderate response, and mean Fatigue score at least 5.0 for at least 8 consecutive weeks for major response. Single response periods and the sum of response periods during 24 months follow-up will be recorded.

SECONDARY OUTCOMES:
Short Form-36 (SF-36) | Changes in SF-36 scores during 24 months follow-up
  SF-36 (ver 1.2) are selfreported by patients at baseline, and at 3, 6, 9, 12, 15, 18, 21 and 24 months follow-up. Changes in Physical health summary score, Physical function, and "Mean of five subdimensions" (Physical function, Bodily pain, Vitality, Social function, General health) are recorded. The difference in course during 24 months follow-up, between the rituximab and placebo groups, will constitute secondary endpoints.
  Also, the difference between rituximab and placebo groups, in changes from baseline to recording at 18 months, for Physical health summary score, Physical function, and "mean of five SF-36 subdimensions", constitute secondary endpoints.
Physical activity (Sensewear armband) | Analyzed at baseline and at interval 17-21 months
  The patients' physical activity level, in a home setting for 7 consecutive days, is recorded using Sensewear armbands, with registration at baseline and repeated in the time interval 17-21 months follow-up. Changes from baseline to analysis during the time interval 17-21 months, for mean number of steps per 24h, maximum number of steps per 24h, mean duration per 24h with activity level at least 3.5 METs, max duration per 24h with activity level at least 3.5 METs, are recorded. The difference between rituximab and placebo groups will constitute secondary endpoints.
Self-recorded "Function level" | Course during 24 months follow-up
  Self-recorded "Function level" (scale 0-100, compared to healthy state, according to a set of examples) are registered every second week. Mean "Function level" for the time intervals 0-4, 4-8, 8-12, 12-16, 16-20, 20-24 months are calculated. The difference in course of "Function level", between the rituximab and placebo groups, constitute a secondary endpoint.
  Also, the differences between the rituximab and placebo groups, for changes in selfreported "Fatigue score" and in selfreported "Function level", calculated from baseline to the mean value during the time interval 16-20 months, constitute secondary endpoints.
Fatigue Severity Scale | 24 months
  Fatigue Severity Scale (FSS) is self-recorded at baseline and at 6, 12, 18, 24 months. The difference between the rituximab and placebo groups, in changes in FSS from baseline to 18 months follow-up, constitutes a secondary endpoint.
Clinical response duration | During 24 months follow-up
  Clinical response periods, defined as consecutive self-recorded Fatigue score at least 4.5 (scale 0-6) for a minimum of 8 weeks, during 24 months follow-up, are recorded.
  The difference in the longest consecutive clinical response period, between rituximab and placebo groups, constitutes a secondary endpoint.
Sustained clinical response at 24 months | Assessment at 24 months
  The difference between rituximab and placebo groups, in fraction of patients with sustained clinical response (defined as Fatigue score of at least 4.5) at 24 months, constitute a secondary endpoint.

OTHER OUTCOMES:
Toxicity and side-effects | During 24 months follow-up
  Toxicity and side effects will be recorded throughout 24 months follow-up, as specified in the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Olav Mella, MD, PhD, Principal Investigator — Dept. of Oncology, Haukeland University Hospital, Bergen, Norway
Locations (5):
- Norway (5):
  - Dept. of Oncology, Haukeland University Hospital, Bergen
  - Notodden Hospital, Notodden
  - CFS/ME centre, Oslo University Hospital, Oslo
  - Division of Rehabilitation Services, University Hospital of North Norway, Tromsø
  - Dept. of Pain and Complex Disorders, St. Olavs Hospital, Trondheim

REFERENCES:
- [Background] Fluge O, Mella O. Clinical impact of B-cell depletion with the anti-CD20 antibody rituximab in chronic fatigue syndrome: a preliminary case series. BMC Neurol. 2009 Jul 1;9:28. doi: 10.1186/1471-2377-9-28. PMID 19566965
- [Background] Fluge O, Bruland O, Risa K, Storstein A, Kristoffersen EK, Sapkota D, Naess H, Dahl O, Nyland H, Mella O. Benefit from B-lymphocyte depletion using the anti-CD20 antibody rituximab in chronic fatigue syndrome. A double-blind and placebo-controlled study. PLoS One. 2011;6(10):e26358. doi: 10.1371/journal.pone.0026358. Epub 2011 Oct 19. PMID 22039471
- [Derived] Fluge O, Rekeland IG, Lien K, Thurmer H, Borchgrevink PC, Schafer C, Sorland K, Assmus J, Ktoridou-Valen I, Herder I, Gotaas ME, Kvammen O, Baranowska KA, Bohnen LMLJ, Martinsen SS, Lonar AE, Solvang AH, Gya AES, Bruland O, Risa K, Alme K, Dahl O, Mella O. B-Lymphocyte Depletion in Patients With Myalgic Encephalomyelitis/Chronic Fatigue Syndrome: A Randomized, Double-Blind, Placebo-Controlled Trial. Ann Intern Med. 2019 May 7;170(9):585-593. doi: 10.7326/M18-1451. Epub 2019 Apr 2. PMID 30934066